CLINICAL TRIAL: NCT01296828
Title: Posture, Tone and Mobility of Lips and Tongue of Mouth Breathing Children
Brief Title: Lips and Tongue of Mouth Breathing Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Marta Assumpção de Andrada e Silva, Pontificia Universidade Catolica de Sao Paulo´s professor
Other Study IDs: CEP PUC/SP 302/2008
Record Dates: First submitted 2011-02-01; First posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2010-11

CONDITIONS: Mouth Breathing
MeSH Terms: conditions — Mouth Breathing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MOUTH BREATHING CHILDREN

SUMMARY:
Purpose: to characterize the posture, tone and mobility of lips and tongue of mouth breathing children.

Methods: 40 mouth breathing children, 26 (65%) male and 14 (35%) female, aging between 7 and 10 years old, were involved in this research realized in São Paulo, SP, Brazil . It was used the MBGR protocol to evaluate the posture, tone and mobility of lips and tongue of mouth breathing children.

ELIGIBILITY:
Inclusion Criteria:

* Mouth breathing children diagnosed by doctor.

Exclusion Criteria:

* Children with mental, neurological or hearing diseases, or with cold or flu at the examination day.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 40 mouth breathing children, 26 (65%) male and 14 (35%) female, aging between 7 and 10 years old, were involved in this research realized in Instituto CEFAC, São Paulo, SP, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Q Marchesan, Study Chair — CEFAC Educação e Saúde
Locations (1):
- Instituto CEFAC, São Paulo, São Paulo, Brazil